CLINICAL TRIAL: NCT05935358
Title: Nuwiq for Perioperative Management Of Patients With Haemophilia A on Emicizumab Regular Prophylaxis Study (NuPOWER)
Brief Title: Nuwiq for Perioperative Management Of Patients With Haemophilia A on Emicizumab Regular Prophylaxis Study
Acronym: NuPOWER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GENA-22
Record Dates: First submitted 2023-06-08; First posted 2023-07-07 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Severe Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nuwiq (Experimental): All patients receiving Nuwiq (recombinant FVIII). Nuwiq will be administered intravenously in accordance with the relevant prescribing information. Treatment will be repeated as necessary every 8-24 hours until adequate wound healing, then - if required - for at least another 7 days to maintain FVIII plasma levels of 30-60 IU/dL.
  Interventions: Drug: Nuwiq

INTERVENTIONS:
Drug: Nuwiq — Nuwiq is a purified B-domain-deleted FVIII glycoprotein synthesised by a genetically engineered human embryonic kidney cell line (HEK 293F).

SUMMARY:
Recombinant factor VIII for the prevention of bleeding in patients with severe haemophilia A undergoing major surgery while receiving emicizumab prophylaxis

DETAILED DESCRIPTION:
Patients with severe haemophilia A receiving emicizumab will often need concomitant FVIII to provide haemostatic cover during major surgery. This prospective, open-label, uncontrolled, single-arm, multinational, multicentre study aims to evaluate the overall perioperative haemostatic efficacy of Nuwiq, a recombinant factor VIII, in combination with emicizumab prophylaxis in male patients over 12 with severe haemophilia A undergoing major surgery.

ELIGIBILITY:
Inclusion Criteria:

* Severe haemophilia A (FVIII activity [FVIII:C] <1%) according to medical history
* Male patients at least 12 years of age
* Previous treatment with any FVIII product(s) for at least 150 exposure days
* On regular prophylaxis with emicizumab for at least 1 month prior to a scheduled major elective surgery requiring FVIII treatment
* Freely given written informed consent of the patient, or parent/legal representative where applicable, obtained in accordance with local regulations

Exclusion Criteria:

* Coagulation disorder other than haemophilia A
* Present or past FVIII inhibitor (≥0.6 Bethesda units [BU]/mL) according to medical history
* Severe liver or kidney disease (alanine aminotransferase [ALT] and/or aspartate aminotransferase [AST] levels >5 times the upper limit of normal; or creatinine >120 μmol/L)
* Known hypersensitivity to Nuwiq's active substance or its excipients (sucrose, sodium chloride, calcium chloride dihydrate, arginine hydrochloride, sodium citrate dihydrate, poloxamer 188)
* Already had surgery in this study
* Current participation in another interventional clinical trial
* Treatment with any investigational medicinal product (IMP) within 30 days prior to screening visit

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Overall haemostatic efficacy | During surgery and until completion of wound healing (e.g. removal of sutures, cessation of drainage, etc.) as defined by the investigator, during the study duration of 30 ± 3 days after the day of surgical procedure
  Overall haemostatic efficacy of treatment measured as binary "success" or "failure". The overall perioperative haemostatic efficacy of Nuwiq will be adjudicated by an Independent Data Monitoring Committee (IDMC) and determined using a composite assessment algorithm that considers the surgeon's assessment of intraoperative haemostatic efficacy and the investigator's assessment of postoperative haemostatic efficacy to classify the overall haemostatic efficacy as success or failure.

SECONDARY OUTCOMES:
Intraoperative haemostatic efficacy | During surgery: From first skin incision to last suture
  Assessment of intraoperative haemostatic efficacy of Nuwiq using a 4-point ordinal scale:
  Excellent: Intraoperative blood loss was lower than or equal to the average expected blood loss for the type of procedure performed in a patient with normal haemostasis and of the same sex, age, and stature
  Good: Intraoperative blood loss was higher than the average expected blood loss but lower or equal to the maximal expected blood loss for the type of procedure in a patient with normal haemostasis.
  Moderate: Intraoperative blood loss was higher than the maximum expected blood loss for the type of procedure performed in a patient with normal haemostasis, but haemostasis was controlled.
  None: Haemostasis was uncontrolled, necessitating a change in the clotting factor replacement regimen.
Postoperative haemostatic efficacy | From end of surgery until completion of wound healing (e.g. removal of sutures, cessation of drainage, etc.) as defined by the investigator, during the study duration of 30 ± 3 days after the day of surgical procedure
  Assessment of postoperative haemostatic efficacy of Nuwiq using a 4-point ordinal scale:
  Excellent: No postoperative bleeding or oozing that was not due to complications of surgery. All postoperative bleeding (due to complications of surgery) was controlled with Nuwiq as anticipated for the type of procedure.
  Good: No postoperative bleeding or oozing that was not due to complications of surgery. Control of postoperative bleeding due to complications of surgery required increased dosing with Nuwiq or additional injections not originally anticipated for the type of procedure.
  Moderate: Some postoperative bleeding and oozing that was not due to complications of surgery. Control of postoperative bleeding required increased dosing with Nuwiq or additional injections not originally anticipated for the type of procedure.
  None: Extensive uncontrolled postoperative bleeding and oozing.
Blood product transfusion levels | From day of surgery until completion of wound healing (e.g. removal of sutures, cessation of drainage, etc.) as defined by the investigator, during the study duration of 30 ± 3 days after the day of surgical procedure
  The number of allogeneic blood products (red blood cells, platelets, and other blood products) transfused
FVIII plasma levels | ≤30 minutes before and 15-30 minutes after Nuwiq injection
  Perioperative plasma levels
Thrombin generation | ≤30 minutes before and 15-30 minutes after Nuwiq injection
  Perioperative thrombin generation
Perioperative haemostatic efficacy per World Federation of Hemophilia (WFH) criteria | Perioperative
  Assessed on WFH recommended 4-point scale:
  Excellent: Intra and post-operative blood loss, with blood component transfusions, similar to non-haemophilic patients. No additional FVIII/bypassing agents Good: Intra/ post-operative blood loss slightly increased over expectation for non-haemophilic patient but clinically insignificant. Blood component transfusions similar to non-haemophilic patient. No additional FVIII/bypassing agents Fair: Intra/ post-operative blood loss increased over expectation for non-haemophilic patients, and additional treatment needed. Extra dose of FVIII/bypassing agents needed or increased blood component of anticipated transfusion requirement Poor: Significant intra- or post-operative blood loss substantially increased over non-haemophilic patient, requires haemophilia-related medical intervention. Unexpected hypotension, transfer to ICU due to bleeding or substantially increased blood component of anticipated transfusion requirement
Thrombotic events | From start of first Nuwiq injection to 30 ± 3 days following the surgical procedure or until day of discharge, whichever is later
  Incidence of thrombotic events during the study
FVIII inhibitor formation | From start of first Nuwiq injection to 30 ± 3 days following the surgical procedure or until day of discharge, whichever is later
  Incidence of FVIII inhibitor formation
Adverse events | From start of first Nuwiq injection to 30 ± 3 days following the surgical procedure or until day of discharge, whichever is later
  Incidence of adverse events recorded during the full study period

CONTACTS AND LOCATIONS:
Overall Officials: Shveta Gupta, MD, Principal Investigator — Arnold Palmer Hospital for Children
Locations (18):
- UT Southwestern Medical Center, Dallas, Texas, United States
- University Hospital Centre Zagreb, Zagreb, Croatia
- Helsinki University Hospital, Helsinki, Finland
- France (2):
  - CHU de Nantes Hôtel-Dieu, Nantes
  - CHRU de Tours, Tours
- Germany (3):
  - Vivantes Klinikum im Friedrichshein (KFH), Berlin
  - Gerinnungszentrum Rhein-Ruhr, Duisburg
  - Universitätsklinikum Hamburg Eppendorf (UKE), Hamburg
- India (2):
  - Christian Medical College Vellore, Vellore, Tamil Nadu
  - St. John's Medical College Hospital, Bengaluru
- Italy (3):
  - Azienda Ospedaliera Pugliese Ciaccio, Catanzaro
  - Azienda Ospedaliero Universitaria Careggi - Centro Emofilia, Florence
  - Centro Trombosi e Malattie Emorragiche, ITCCS Humanitas Research Hospital, Milan
- Centre for Haemopilia, Institute for transfusion medicine of Republic of North Macedonia, Skopje, North Macedonia
- Clinical Center for Serbia Belgrade, Belgrade, Serbia
- Spain (2):
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- St. James's University Hospital, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srivastava A, Kanny A, Langer F, Kubicek-Hofmann C, Alvarez Roman MT, Nunez Vazquez R, Boban A, Dejanova-Ilijevska V, Miljic P, Garcia J, Halimeh S, Drillaud N, Valentin JB, Mancuso ME, Castaman G, Santoro RC, Lehtinen AE, Abraham A, Hashimoto M, Knaub S. NuPOWER (Nuwiq for Perioperative management Of patients With haemophilia A on Emicizumab Regular prophylaxis): protocol for an open-label, single-arm, multicentre study. BMJ Open. 2025 Oct 28;15(10):e102657. doi: 10.1136/bmjopen-2025-102657. PMID 41151952